CLINICAL TRIAL: NCT02282891
Title: A Randomized-Controlled Trial to Compare the Effect of Propofol vs. "Ketofol" on Hemodynamic Stability During Induction of General Anesthesia
Brief Title: Compare the Effect of Propofol vs. "Ketofol" on Hemodynamic Stability During Induction of General Anesthesia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were ever recruited and enrolled.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1406014189
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Patients With "ASA 3" Designation
Keywords: propofol; ketofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Induction of general Anesthesia using propofol 2mg/kg
  Interventions: Drug: Propofol
- Propofol/Ketamine (ketofol) (Experimental): Induction of general anesthesia using a mixture of 1.5mg/kg:0.75mg/kg Propofol/ketamine
  Interventions: Drug: Propofol-Ketamine

INTERVENTIONS:
Drug: Propofol — Induction of general anesthesia using propofol 2mg/kg
  Other Names: Diprivan
  Arms: Propofol
Drug: Propofol-Ketamine — Induction of general anesthesia using a mixture of 1.5 mg/kg:0.75 mg/kg propofol/ketamine
  Other Names: ketofol
  Arms: Propofol/Ketamine (ketofol)

SUMMARY:
The purpose of this study is to compare the hemodynamic effects of a standardized induction of general anesthesia with either propofol or ketofol in patients with physical status classification ASA 3. The study will be a double blinded, randomized controlled trial (RCT) with two arms of treatment groups. One arm will consist of induction of general anesthesia using a mixture of 1.5mg/kg:0.75mg/kg Propofol/ketamine (ketofol) and the induction dose will be 1.5mg/kg of propofol and 0.75mg/kg of ketamine; the second arm will consist of induction of general anesthesia using propofol 2mg/kg. The primary outcome of the intervention will consist of hemodynamic changes during the first 30 minutes after induction of general anesthesia.

DETAILED DESCRIPTION:
The anesthetic agent propofol can result in hypotension when used for induction of general anesthesia. Recent trials suggest that even a short duration of hypotension during induction of anesthesia can adversely affect organ function and overall outcome.1 To overcome the hypotensive effect of propofol, ketamine, which has sympathomimetic effects, has been combined with propofol to produce a mixture labeled "ketofol", which has been used both for procedural sedation and induction of general anesthesia. Clinical trials have shown that ketofol can attenuate the hypotensive effects of propofol during procedural sedation or induction of general anesthesia in patients whose physical status is 1 or 2 according to the American Society of Anesthesiologists (ASA 1-2), i.e., healthy patients or those with mild-moderate systemic illness.2,3 Clinically, it is important to demonstrate the efficacy of ketofol in attenuating hypotensive effects of propofol in sicker patients, i.e., patients with physical status ASA 3. The purpose of this study is to compare the hemodynamic effects of a standardized induction of general anesthesia with either propofol or ketofol in patients with physical status classification ASA 3. The study will be a double blinded, randomized controlled trial (RCT) with two arms of treatment groups. One arm will consist of induction of general anesthesia using a mixture of 1.5mg/kg:0.75mg/kg Propofol/ketamine (ketofol) and the induction dose will be 1.5mg/kg of propfol and 0.75mg/kg of ketamine; the second arm will consist of induction of general anesthesia using propofol 2mg/kg. The primary outcome of the intervention will consist of hemodynamic changes during the first 30 minutes after induction of general anesthesia.

Baseline demographics collected for each patient will include:

1. age
2. sex
3. ASA physical status
4. Hx of HTN
5. Hx of PONV
6. Preoperative pain score

The standardized induction of anesthesia will consist of intravenous administration of midazolam 0.04mg/kg, lidocaine 1 mg/kg, fentanyl 1-2 mcg/kg, glycopyrrolate 0.004 mg/kg, an unlabeled pre-prepared, covered syringe which will be prepared by the Yale Anesthesia satellite pharmacist containing either propofol 2mg/kg or a mixture propofol 1.5mg/kg and ketamine 0.75mg/kg, the amount of which will be pre-determined based on the patient weight, and rocuronium 0.6 mg/kg. A backup 10cc syringe of the study drug will be available as well if the initial dose is inadequate. The choice of propofol and ketamine dosing is based on a study cited earlier by Smischney et al in 2012 that addresses ASA 1-2 patients undergoing induction of general anesthesia. Endotracheal intubation will take place after adequate muscle relaxation has been determined using fade of train of four on a nerve stimulator placed over the ulnar nerve. Additional medication to facilitate induction will be used according to the judgment of the anesthesia provider with a backup syringe of the same study drug. Inhalational anesthesia will be administered after confirmation of endotracheal intubation. Treatment of hypotension will be according to the anesthesia provider. Amounts of intravenous fluids as well as doses of vasopressor that are used during induction and in the subsequent 30 minutes after endotracheal intubation will be obtained from the anesthesia record.

The first blood pressure (BP) upon arrival to the operating room before any anesthetic medications are administered will be the reference (baseline) blood pressure. BP will be measured every 1 minute from one minute before induction until 30 minutes after endotracheal intubation.

The primary outcome of the study will be the number of time points during which the blood pressure was below 20% of the baseline BP. Secondary outcomes will include:

1. Severity of hypotension as determined by the gradient of each blood pressure measurement from the baseline BP.
2. The total dosage of vasopressors administered during induction and up to 30 minutes after endotracheal intubation
3. The total amount of IV fluids administered during induction and up to 30 minutes after endotracheal intubation.
4. The total amount of additional medications used during induction and up to 30 minutes after endotracheal intubation.
5. Total intraoperative as well as postoperative opioid dosage used.
6. Presence or absence of PONV and severity
7. Intraoperative prophylaxis and postoperative treatment of PONV

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-80 scheduled for elective surgery
* Physical status ASA 3.

Exclusion Criteria:

* Patients with a physical status of ASA 1,2, 4 or 5,
* Prior adverse reaction to propofol, ketamine or both

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of time points during which blood pressure was below 20% of baseline BP | up to 30 minutes after intubation
  The number of time points during which the blood pressure was below 20% of the baseline BP. The first blood pressure upon arrival to the operating room before any anesthetic medications are administered will be the reference (baseline) blood pressure. BP will be measured every 1 minute from one minute before induction until 30 minutes after endotracheal intubation.

SECONDARY OUTCOMES:
Severity of hypotension | up to 30 minutes after intubation
  As determined by the gradient of each blood pressure measurement from the baseline BP
Total dosage of vasopressors administered | up to 30 minutes after intubation
  The total dosage of vasopressors administered during induction and up to 30 minutes after endotracheal intubation
Amount of IV fluids administered | up to 30 minutes after intubation
  The total amount of IV fluids administered during induction and up to 30 minutes after endotracheal intubation.
Additional Medication Usage | up to 30 minutes after intubation
  The total amount of additional medications used during induction and up to 30 minutes after endotracheal intubation.
Total Opioid Dosage Used | up to 30 minutes after intubation
  Total intraoperative as well as postoperative opioid dosage used.
Post Operative Nausea and Vomiting (PONV) Severity | 72 hours post surgery
  Presence or absence of PONV and severity within 72 hours of surgery
Treatment of Post Operative Nausea and Vomiting (PONV) | 72 hours post surgery
  Number and dose of anti-emetics given within 72 hours of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jamel P Ortoleva, MD, Principal Investigator — Yale University; Jean Charchaflieh, MD,MPH,DrPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States